CLINICAL TRIAL: NCT04140084
Title: Wiki Head CT Choice Study: Adaptation of Two Decision Aids to Support Shared Decision Making About Performing a Head CT for Adult and Pediatric Victims of Mild Traumatic Brain Injury
Brief Title: Wiki Head CT Choice Study: Adaptation of US Two Decision Aids to a Québec Local Context
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Archambault, Associate Professor, Laval University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-393 - WikiDécisionTDM
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Mild Traumatic Brain Injury; Emergencies; Decision-making
Keywords: Emergency Department; Mild Traumatic Brain Injury; Shared decision-making; Decision aids; Head computed tomography
MeSH Terms: conditions — Brain Concussion; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Translation, Redesign and Rapid prototyping with clinicians (No Intervention): This step includes a translation of the tools (English to French) and a redesign work of the original tools. Then, the study will include clinicians (at least 20) from two healthcare settings (CHU Sainte-Justine, and the CISSS-CA (Hotel-Dieu de Levis). After a presentation of the two tools during the Emergency Physicians' departmental meetings, the written comments about the prototype version will be collected. A revision of the prototypes is scheduled at the end of this step.
- Rapid prototyping with patients (No Intervention): This step will include the assessment of the tools by patients (or parents of patients) that have had a previous mTBI at the CISSS-CA (Hotel-Dieu de Levis). The comments about the adult and pediatric prototypes (5 adult patients, 5 parents of pediatric patients) will be collected through interviews. A revision of the prototypes is scheduled at the end of this step.
- Real-life clinical meetings (Experimental): This step will include a presentation of the tools to 5 emergency physicians so that they can use the tools with patients (5 adults, 5 parents of pediatric patients) in a realistic setting to identify any problems of use. The clinicians and patients that had used the tools during the clinical encounters will be then met during cognitive interviews to collect their comments on the tools and to address any usability issues. A final revision of the prototypes is scheduled at the end of this step.
  Interventions: Device: Real-life clinical meetings
- Training session developement (No Intervention): This step includes the development of a training session on how to perform SDM with patients facing the decision to undergo head CTs for mTBI and about how to use our newly developed decision aids in this clinical setting. The content of the training session will be adapted to the needs, goals, strengths and limitations observed during the focus groups (departmental meetings) exploring health professionals' barriers to using a decision aid about head CTs in mTBI. The expertise of SAVIE (www.savie.ca) in producing online and interactive elearning programs will be mobilized in order to produce a training program that will integrate the content the investigators will have identified as the main skills, knowledge and competencies needing development among our health professionals to stimulate the use of SDM and our decision aids. SAVIE will produce a virtual elearning program adaptable to all media (PC, mobile device, tablet) and different health professionals.
- Retrospective analysis (No Intervention): This step will retrospectively analyze the medical records of traumatic brain injury adult patients (adult, 350, Hotel-Dieu de Levis) and pediatric patients (406, CHU de Sainte-Justine and Hotel-Dieu de Levis)) randomly selected throughout the year preceding this study in each of the two centers to determine the rate of head CT ordering, the head CT result and the appropriateness of having ordered the head CT based on the CCHR and PECARN criteria. One reviewer will judge the appropriateness of having done a CT scan according to the CCHR and PECARN criteria based on a structured extraction form that will previously be approved by the study's steering committee. To ensure validity, 10% of the analysis will be reviewed by an expert. The reviewer will look at prehospital data collection, triage information, physician's notes, nursing notes and head CT requisition form information to determine if any of the clinical decision rule criteria are present.

INTERVENTIONS:
Device: Real-life clinical meetings — Study coordinators will identify potentially eligible parent/patient dyads and adult patients based on a chief complaint related to head trauma recorded at the time of ED registration and communication with treating clinicians in realtime. After using the decision aid with their health professional, a cognitive interview session will then be organized with the dyads of participants (parents/patients and clinicians) to address any usability issues. These interviews will be audio recorded and transcribed verbatim for content analysis and future reference. This process will allow to identify any conceptual barriers and unanticipated user needs. Written consent form will be signed by participants.
  Arms: Real-life clinical meetings

SUMMARY:
This study aims to adapt two decision aids (DAs) (pediatric and adult) developed in the United States to the Quebec context to develop context-adapted tools and training program that will facilitate the process of shared decision-making while taking a decision to use head computed tomography (CT scan) with patients suffering from a mild traumatic brain injury.

DETAILED DESCRIPTION:
Background: Mild traumatic brain injury (mTBI) is among the most common neurological conditions with an estimated annual incidence rate of 450 to 650/100,000 in Canada. Head computed tomography (CT) scans are used as the reference standard test to rule out life-threatening complications, such as intracranial hemorrhage, but present potential exposition risks for the patient. Despite the use of clinical decision rules (Canadian Head CT Rule; Pediatric Head Injury/Trauma Algorithm (PECARN)), head CTs remain overused. Two decision aids (pediatric and adult) developed in the United States (U.S.) may help reduce the use of CTs for mTBI.

The goal of this study is to address the challenges of adapting two existing decision aids to local contexts. Stakeholders, including patients, or parents of patients, will be involved in adapting and validating the two existing decision aids to a local context and to create a training program about shared decision-making (SDM) in trauma care.

Objectives:

1. Translate two decision aids for head CTs (pediatric and adult) developed in the United States and adapt them to the Quebec context;
2. Create training for Emergency Medicine professionals on adopting decision aids with mTBI patients;
3. Measure the appropriate use of CTs in two hospitals(CHU de Sainte-Justine, Hotel-Dieu de Levis) before implementing the tools.

Methods:

Phase 1 will be the translation and adaptation of two decision aids to support decision-making about performing a head CT for adult and pediatric mTBI using an iterative user-centered approach. (Translation of the decision aids on the use of CT scans for mTBI (pediatric and adult) produced in the United States; simple ethnographic observation of the interactions of emergency health professionals and mTBI patients to understand the needs of patients, family members and health professionals in deciding to conduct a head CT for mTBI patients for the redesign of the tools; rapid prototyping of our different decision aids using interviews and real-life clinical encounters.)

Phase 2 will be the development of a training session for healthcare professionals.

Phase 3 will be a retrospective analysis of medical records to evaluate the use of head CT for mTBI patients in two hospitals (pediatric and adult).

Expected results:

This study will adapt two decision aids to the context of trauma care in Quebec and create a training program about shared decision-making and decision aids in the context of the care of mTBI patients. The final content and user interface of the decision aid/training session will be influenced by the multiple comments received from the participants in this study. This novel online and in -person training program will be instrumental in implementing our novel decision aid in practice. The results generated from the implementation of the intervention will help other centers in Quebec, Canada and abroad use the educational program and decision aid. The results of this research project will contribute to the enhancement of many research fields such as the involvement of end- users in the development process of decision aids. This research project will offer new learning opportunities for graduate students to study how collaboration among multiple stakeholders can improve patient outcomes and how to develop patient- centered tools that respond to their needs and those of the clinicians that care for them. Finally, this project will advance our understanding of the use of shared decision-making and decision aids in the field of trauma care.

ELIGIBILITY:
Rapid-prototyping steps:

Inclusion criteria:

* For the pediatric decision aid: Parents seeking care for a child or an adolescent that are less than 18 years old. The child must have experienced blunt head trauma (above the eyebrows and not isolated to face or eyes).The child must have at least one of the PECARN risk factors for clinically important TBI (except for the two higher risk variables of altered mental status or signs of skull fracture).
* For the adult decision aid: Adult participants that have had a diagnosis of mTBI before the interview or having a mTBI to be diagnosed by the physician at the moment and needs to make a decision about having a CTs.
* Eligible clinicians will be attending physicians, fellows, and residents caring for children or adult with minor head trauma.

Exclusion criteria:

* For the pediatric decision aid: Suspected case of child abuse.
* For the adult decision aid: No exclusion criteria.

Retrospective analysis:

Inclusion criteria:

* Children that have experienced blunt head trauma (above the eyebrows and not isolated to face or eyes).
* Children that have at least one of the PECARN risk factors for clinically important TBI (except for the two higher risk variables of altered mental status or signs of skull fracture).
* Adults who have experienced blunt head trauma (above the eyebrows and not isolated to face or eyes) within 24 hours without any of the high risk or medium risk CCHR criteria that mandate performing a head CT.

Exclusion criteria:

* Children with signs of skull fracture, GCS < 15 or other signs of altered mental status, brain tumour, penetrating head trauma, bleeding disorder or coagulopathy, ventricular shunt, preexisting neurological disease, syncope or seizure that preceded the head trauma, transferred to the ED with imaging already obtained, known pregnancy, suspected abuse, or > 2 PECARN risk factors.
* Adults that have a Glasgow coma scale less than 13, an obvious open skull fracture, take oral anticoagulants, or antiplatelet agents (excluding aspirin), or have a bleeding disorder, no causal factor of trauma (i.e. epilepsy, cardiac arrest), pregnancy, came back to emergency for the same head injury, no symptoms of head injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Adapting two decision aids to the context of trauma care in Quebec. | interviews or departmental meeting or clinical encounters with participants over a duration of one year
  Adapting two decision aids to the context of trauma care in Quebec using interviews of 5 adult patients and 5 parents of pediatric patients and 2 focus group (during departmental meeting), as well as real-life medical encounters with 5 adult patients and 5 pediatric patients (and parents).
Create a training program about SDM in the context of the care of mTBI patients. | meetings over a 3 months periods
  Create a training program about SDM in the context of the care of mTBI patients with specialists using the data and comments gathered during the rapid prototyping phase.
Understand CT scan overuse in two hospitals. | retrospective analysis during a year (10 hours/week)
  Understand CT scan overuse in two hospitals, one pediatric and one general hospital, by looking at health records (randomized samples).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre integre de sante et de services sociaux de Chaudiere-Appalaches, Lévis, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abras, Chadia, Diane Maloney-Krichmar, and Jenny Preece. 2004. "User-Centered Design." Bainbridge, W. Encyclopedia of Human-Computer Interaction. Thousand Oaks: Sage Publications 37 (4): 445-56.
- [Background] Legare F, O'Connor AM, Graham ID, Wells GA, Tremblay S. Impact of the Ottawa Decision Support Framework on the agreement and the difference between patients' and physicians' decisional conflict. Med Decis Making. 2006 Jul-Aug;26(4):373-90. doi: 10.1177/0272989X06290492. PMID 16855126
- [Background] Archambault PM, van de Belt TH, Grajales FJ 3rd, Faber MJ, Kuziemsky CE, Gagnon S, Bilodeau A, Rioux S, Nelen WL, Gagnon MP, Turgeon AF, Aubin K, Gold I, Poitras J, Eysenbach G, Kremer JA, Legare F. Wikis and collaborative writing applications in health care: a scoping review. J Med Internet Res. 2013 Oct 8;15(10):e210. doi: 10.2196/jmir.2787. PMID 24103318
- [Background] Archambault PM. WikiBuild: a new application to support patient and health care professional involvement in the development of patient support tools. J Med Internet Res. 2011 Dec 8;13(4):e114. doi: 10.2196/jmir.1961. PMID 22155746
- [Background] Archambault PM, Bilodeau A, Gagnon MP, Aubin K, Lavoie A, Lapointe J, Poitras J, Croteau S, Pham-Dinh M, Legare F. Health care professionals' beliefs about using wiki-based reminders to promote best practices in trauma care. J Med Internet Res. 2012 Apr 19;14(2):e49. doi: 10.2196/jmir.1983. PMID 22515985
- [Background] Archambault PM, Gagnon S, Gagnon MP, Turcotte S, Lapointe J, Fleet R, Cote M, Beaupre P, Le Sage N, Emond M, Legare F. Development and validation of questionnaires exploring health care professionals' intention to use wiki-based reminders to promote best practices in trauma. JMIR Res Protoc. 2014 Oct 3;3(3):e50. doi: 10.2196/resprot.3762. PMID 25281856
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] "Choosing Wisely Canada." n.d. Choosing Wisely Canada. Five Things Physicians and Patients Should Question. Accessed June 2, 2015. http://www.choosingwiselycanada.org/recommendations/emergencymedicine/.
- [Background] Curran JA, Brehaut J, Patey AM, Osmond M, Stiell I, Grimshaw JM. Understanding the Canadian adult CT head rule trial: use of the theoretical domains framework for process evaluation. Implement Sci. 2013 Feb 21;8:25. doi: 10.1186/1748-5908-8-25. PMID 23433082
- [Background] Dis, Iso. 2009. "9241-210: 2010. Ergonomics of Human System Interaction-Part 210: Human- Centred Design for Interactive Systems." International Standardization Organization (ISO). Switzerland.
- [Background] Evans R, Edwards A, Brett J, Bradburn M, Watson E, Austoker J, Elwyn G. Reduction in uptake of PSA tests following decision aids: systematic review of current aids and their evaluations. Patient Educ Couns. 2005 Jul;58(1):13-26. doi: 10.1016/j.pec.2004.06.009. PMID 15950832
- [Background] Flynn D, Knoedler MA, Hess EP, Murad MH, Erwin PJ, Montori VM, Thomson RG. Engaging patients in health care decisions in the emergency department through shared decision-making: a systematic review. Acad Emerg Med. 2012 Aug;19(8):959-67. doi: 10.1111/j.1553-2712.2012.01414.x. Epub 2012 Jul 31. PMID 22853804
- [Background] Gagliardi AR, Alhabib S; members of Guidelines International Network Implementation Working Group. Trends in guideline implementation: a scoping systematic review. Implement Sci. 2015 Apr 21;10:54. doi: 10.1186/s13012-015-0247-8. PMID 25895908
- [Background] Gagliardi AR, Brouwers MC, Bhattacharyya OK. The development of guideline implementation tools: a qualitative study. CMAJ Open. 2015 Jan 13;3(1):E127-33. doi: 10.9778/cmajo.20140064. eCollection 2015 Jan-Mar. PMID 25844365
- [Background] Garrett, Jesse James. 2010. The Elements of User Experience: User-Centered Design for the Web and Beyond. Pearson Education.
- [Background] Gould, John D., and Clayton Lewis. 1985. "Designing for Usability: Key Principles and What Designers Think." Communications of the ACM 28 (3): 300-311.
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Greenhalgh T, Howick J, Maskrey N; Evidence Based Medicine Renaissance Group. Evidence based medicine: a movement in crisis? BMJ. 2014 Jun 13;348:g3725. doi: 10.1136/bmj.g3725. PMID 24927763
- [Background] Grilli R, Lomas J. Evaluating the message: the relationship between compliance rate and the subject of a practice guideline. Med Care. 1994 Mar;32(3):202-13. doi: 10.1097/00005650-199403000-00002. PMID 8145598
- [Background] Gurses AP, Ozok AA, Pronovost PJ. Time to accelerate integration of human factors and ergonomics in patient safety. BMJ Qual Saf. 2012 Apr;21(4):347-51. doi: 10.1136/bmjqs-2011-000421. Epub 2011 Nov 30. PMID 22129929
- [Background] Gvero, Igor. 2013. "Observing the User Experience, 2nd Edition: A Practitioner's Guide to User Research by Elizabeth Goodman, Mike Kuniavsky, and Andrea Moed." ACM SIGSOFT Software Engineering Notes 38 (2): 35-35.
- [Background] Hess EP, Grudzen CR, Thomson R, Raja AS, Carpenter CR. Shared Decision-making in the Emergency Department: Respecting Patient Autonomy When Seconds Count. Acad Emerg Med. 2015 Jul;22(7):856-64. doi: 10.1111/acem.12703. Epub 2015 Jun 25. PMID 26112797
- [Background] Hess EP, Wyatt KD, Kharbanda AB, Louie JP, Dayan PS, Tzimenatos L, Wootton-Gorges SL, Homme JL, Pencille R N L, LeBlanc A, Westphal JJ, Shepel K, Shah ND, Branda M, Herrin J, Montori VM, Kuppermann N. Effectiveness of the head CT choice decision aid in parents of children with minor head trauma: study protocol for a multicenter randomized trial. Trials. 2014 Jun 25;15:253. doi: 10.1186/1745-6215-15-253. PMID 24965659
- [Background] Krejcie, Robert V., and Daryle W. Morgan. 1970. "Determining Sample Size for Research Activities." Educational and Psychological Measurement 30 (3): 607-10.
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Background] Legare F, Labrecque M, Cauchon M, Castel J, Turcotte S, Grimshaw J. Training family physicians in shared decision-making to reduce the overuse of antibiotics in acute respiratory infections: a cluster randomized trial. CMAJ. 2012 Sep 18;184(13):E726-34. doi: 10.1503/cmaj.120568. Epub 2012 Jul 30. PMID 22847969
- [Background] Legare F, Ratte S, Stacey D, Kryworuchko J, Gravel K, Graham ID, Turcotte S. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2010 May 12;(5):CD006732. doi: 10.1002/14651858.CD006732.pub2. PMID 20464744
- [Background] Liabsuetrakul T, Chongsuvivatwong V, Lumbiganon P, Lindmark G. Obstetricians' attitudes, subjective norms, perceived controls, and intentions on antibiotic prophylaxis in caesarean section. Soc Sci Med. 2003 Nov;57(9):1665-74. doi: 10.1016/s0277-9536(02)00550-6. PMID 12948575
- [Background] Mao, Ji-Ye, Karel Vredenburg, Paul W. Smith, and Tom Carey. 2005. "The State of User- Centered Design Practice." Communications of the ACM 48 (3): 105-9.
- [Background] Mathews JD, Forsythe AV, Brady Z, Butler MW, Goergen SK, Byrnes GB, Giles GG, Wallace AB, Anderson PR, Guiver TA, McGale P, Cain TM, Dowty JG, Bickerstaffe AC, Darby SC. Cancer risk in 680,000 people exposed to computed tomography scans in childhood or adolescence: data linkage study of 11 million Australians. BMJ. 2013 May 21;346:f2360. doi: 10.1136/bmj.f2360. PMID 23694687
- [Background] McKillop A, Crisp J, Walsh K. Practice guidelines need to address the 'how' and the 'what' of implementation. Prim Health Care Res Dev. 2012 Jan;13(1):48-59. doi: 10.1017/S1463423611000405. Epub 2011 Oct 13. PMID 22008308
- [Background] Melnick ER, Lopez K, Hess EP, Abujarad F, Brandt CA, Shiffman RN, Post LA. Back to the Bedside: Developing a Bedside Aid for Concussion and Brain Injury Decisions in the Emergency Department. EGEMS (Wash DC). 2015 Jun 29;3(2):1136. doi: 10.13063/2327-9214.1136. eCollection 2015. PMID 26290885
- [Background] Munro S, Stacey D, Lewis KB, Bansback N. Choosing treatment and screening options congruent with values: Do decision aids help? Sub-analysis of a systematic review. Patient Educ Couns. 2016 Apr;99(4):491-500. doi: 10.1016/j.pec.2015.10.026. Epub 2015 Nov 2. PMID 26549169
- [Background] O'Connor, A. M., D. Stacey, and M. J. Jacobsen. 2014. "Ottawa Decision Support Tutorial: Improving Practitioners' Decision Support Skills Ottawa Hospital Research Institute: Patient Decision Aids; 2011." Disponible En Ligne: Https://decisionaid. Ohri. ca/ODST/pdfs/ODST. Pdf.
- [Background] O'Connor AM, Tugwell P, Wells GA, Elmslie T, Jolly E, Hollingworth G, McPherson R, Bunn H, Graham I, Drake E. A decision aid for women considering hormone therapy after menopause: decision support framework and evaluation. Patient Educ Couns. 1998 Mar;33(3):267-79. doi: 10.1016/s0738-3991(98)00026-3. PMID 9731164
- [Background] O'Connor AM, Bennett CL, Stacey D, Barry M, Col NF, Eden KB, Entwistle VA, Fiset V, Holmes-Rovner M, Khangura S, Llewellyn-Thomas H, Rovner D. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD001431. doi: 10.1002/14651858.CD001431.pub2. PMID 19588325
- [Background] Parachute. 2015. "The Cost of Injury in Canada." Toronto, Ontario.
- [Background] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Background] Pronovost PJ. Enhancing physicians' use of clinical guidelines. JAMA. 2013 Dec 18;310(23):2501-2. doi: 10.1001/jama.2013.281334. No abstract available. PMID 24310916
- [Background] Quine, Lyn. 2002. "Social Cognition Models and Changing Health Behaviours." Changing Health Behaviour, 1.
- [Background] Rodham K, Gavin J, Coulson N, Watts L. Co-creation of information leaflets to meet the support needs of people living with complex regional pain syndrome (CRPS) through innovative use of wiki technology. Inform Health Soc Care. 2016;41(3):325-39. doi: 10.3109/17538157.2015.1008491. Epub 2015 Feb 24. PMID 25710714
- [Background] Ryu WH, Feinstein A, Colantonio A, Streiner DL, Dawson DR. Early identification and incidence of mild TBI in Ontario. Can J Neurol Sci. 2009 Jul;36(4):429-35. doi: 10.1017/s0317167100007745. PMID 19650352
- [Background] Schaeffer, M., and B. J. Moore. 2012. "User-Centered Design: Clothing the EMR Emperor." In Proceedings of the 2012 Symposium on Human Factors and Ergonomics in Health Care: Human Factors and Ergonomics Society, 166-72. Citeseer.
- [Background] Shneiderman, Ben. 2010. Designing the User Interface: Strategies for Effective Human- Computer Interaction. Pearson Education India.
- [Background] Standardization, I. O. F. 2010. "Ergonomics of Human-System Interaction: Part 210: Human- Centred Design for Interactive Systems." ISO.
- [Background] Stiell IG, Bennett C. Implementation of clinical decision rules in the emergency department. Acad Emerg Med. 2007 Nov;14(11):955-9. doi: 10.1197/j.aem.2007.06.039. Epub 2007 Oct 8. PMID 17923717
- [Background] Stiell IG, Clement CM, Rowe BH, Schull MJ, Brison R, Cass D, Eisenhauer MA, McKnight RD, Bandiera G, Holroyd B, Lee JS, Dreyer J, Worthington JR, Reardon M, Greenberg G, Lesiuk H, MacPhail I, Wells GA. Comparison of the Canadian CT Head Rule and the New Orleans Criteria in patients with minor head injury. JAMA. 2005 Sep 28;294(12):1511-8. doi: 10.1001/jama.294.12.1511. PMID 16189364
- [Background] Stiell IG, Wells GA, Vandemheen K, Laupacis A, Brison R, Eisenhauer MA, Greenberg GH, MacPhail I, McKnight RD, Reardon M, Verbeek R, Worthington J, Lesiuk H. Variation in ED use of computed tomography for patients with minor head injury. Ann Emerg Med. 1997 Jul;30(1):14-22. doi: 10.1016/s0196-0644(97)70104-5. PMID 9209219
- [Background] Straus, Sharon, Jacqueline Tetroe, and Ian D. Graham. 2013. Knowledge Translation in Health Care: Moving from Evidence to Practice. John Wiley & Sons.
- [Background] Tesch, Renata. 1990. Qualitative Research: Analysis Types and Software Tools. Psychology Press.
- [Background] Van De Belt, Tom H. 2011. "Wikis as an Opportunity to Improve Patient Participation in Developing Information Leaflets: A Demonstration Project in Infertility Patients." In Medicine 2.0 Conference. JMIR Publications Inc., Toronto, Canada. http://www.medicine20congress.com/ocs/index.php/med/med2011/paper/view/582.
- [Background] Vilar, Polona. 2010. "Designing the User Interface: Strategies for Effective Human-Computer Interaction (5th Edition)." Journal of the American Society for Information Science. American Society for Information Science 61 (5): 1073-74.
- [Background] Virzi, Robert A. 1992. "Refining the Test Phase of Usability Evaluation: How Many Subjects Is Enough?" Human Factors 34 (4): 457-68.
- [Background] Witteman HO, Dansokho SC, Colquhoun H, Coulter A, Dugas M, Fagerlin A, Giguere AM, Glouberman S, Haslett L, Hoffman A, Ivers N, Legare F, Legare J, Levin C, Lopez K, Montori VM, Provencher T, Renaud JS, Sparling K, Stacey D, Vaisson G, Volk RJ, Witteman W. User-centered design and the development of patient decision aids: protocol for a systematic review. Syst Rev. 2015 Jan 26;4(1):11. doi: 10.1186/2046-4053-4-11. PMID 25623074